CLINICAL TRIAL: NCT06244576
Title: Emotional Dysregulation and Maladaptive Overcontrol in Anorexia Nervosa and the Effect of Radically Open Dialectical Behaviour Therapy
Brief Title: Emotional Dysregulation, Maladaptive Overcontrol in Anorexia - Effect of Radically Open Dialectical Behaviour Therapy
Acronym: EMARO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 278846
Record Dates: First submitted 2024-01-22; First posted 2024-02-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-02

CONDITIONS: Anorexia Nervosa; Anorexia in Adolescence; Anorexia Nervosa, Atypical
Keywords: Anorexia nervosa; Intervention; Multiple baseline case-series experimental design study; Primary outcome: EDE-Q total score; RO DBT; Feasibility
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radically Open Dialectical Behaviour Therapy (RO-DBT) (Experimental): RO-DBT consists of a 1 hour weekly individual session and a 2,5 hour weekly group skill training during 32 weeks in accordance with the published treatment manual and session guides for RO-DBT. For skills training, the 31 patients will be divided into four equal groups in terms on number.
  Interventions: Behavioral: Radically Open Dialectical Behaviour Therapy (RO-DBT)

INTERVENTIONS:
Behavioral: Radically Open Dialectical Behaviour Therapy (RO-DBT) — RO-DBT is a trans diagnostic intervention specifically designed to treat a spectrum of disorders characterized by excessive overcontrol such as anorexia nervosa, autism spectrum disorder, refractory depression, cluster c personality disorders, and mood disorders.

SUMMARY:
This clinical trial employs a two-fold approach, utilizing a single-arm feasibility design within a larger multiple baseline experimental case series study framework over 32 weeks. The study aims to investigate both the feasibility and efficacy of Radically Open Dialectical Behaviour Therapy (RO-DBT) in patients with anorexia nervosa (AN). Feasibility will be assessed through treatment retention, data collection engagement, patient satisfaction, and the occurrence of adverse events. Efficacy outcomes will focus on RO-DBT's impact on ED psychopathology, obsessive-compulsive personality traits, EDR, and BMI.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is characterized by high chronicity and mortality rates. Despite its relatively high prevalence, effective treatments remain elusive, often resulting in extended treatment durations and high dropout rates. Emotional dysregulation (EDR) and obsessive-compulsive personality traits are central to the psychopathology of AN, directly contributing to the disorder's severity and persistence. Radically Open Dialectical Behaviour Therapy (RO-DBT) targets the psychopathology mentioned above and has shown promise in pilot studies with AN patients.

Given the urgent need for effective AN treatments and the potential of RO-DBT, this study aims to investigate both the feasibility and efficacy of this therapy in a clinical setting. The study will employ a single-arm feasibility design within a multiple baseline experimental case series framework over 32 weeks, involving 31 patients aged 16 years and older diagnosed with typical or atypical AN. All assessments will utilize validated psychometric instruments, and trained psychotherapists will administer RO-DBT.

Feasibility will be assessed through:

* Treatment retention
* Data collection engagement
* Patient satisfaction with treatment
* Occurrence of adverse events.

The primary efficacy outcome this trial aims to investigate is:

* Does RO-DBT reduce eating disorder psychopathology in AN as measured by the Eating Disorder Examination Questionnaire (EDE-Q)?

The secondary efficacy outcomes this trial aims to investigate are:

* Does RO-DBT reduce emotional dysregulation in AN as measured by change in the Expressive Suppression subscore of Emotion Regulation Questionnaire (ERQ)?
* Does RO-DBT reduce obsessive-compulsive personality traits in AN as measured by change in the total score of the Five-Factor Obsessive Compulsive Inventory (FFOCI-SF)
* Does RO-DBT increase body weight as measured by change in Body Mass Index (BMI)?

We hypothesize that RO-DBT will be a feasible treatment option for individuals with AN. Furthermore, we anticipate observing reductions in ED psychopathology and expressive suppression, alongside an increase in BMI, between pre- and post-treatment assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of anorexia nervosa or atypical nervosa (i.e., in partial remission with a BMI above ~18.5 but meets criteria B and/or C) according to the Diagnostic and Statistical Manual fifth edition (DSM-5)
* Signed written informed consent form
* Age 16-65
* Sufficient knowledge of Swedish

Exclusion Criteria:

* Substance dependence
* Not willing to accept randomization
* Undergoing simultaneous psychotherapy via another healthcare provider
* Intellectual disability
* Any psychiatric, medical or social condition whether or not listed above, due to which, in the judgment of the investigators and after any consults if indicated, participation in the study is not in the best interest of the patient.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The Eating Disorder Examination Questionnaire (EDE-Q) | 32 weeks
  A 36-item self-report questionnaire designed to measure eating disorder symptoms. The range of scores is 0-132. Higher scores mean more eating disorder symptoms

SECONDARY OUTCOMES:
The Five Factor Obsessive Compulsive Inventory - Short Form (FFOCI-SF) | 32 weeks
  A 48-item self-report questionnaire designed to measure obsessive-compulsive personality traits. The range of scores is 48-240. Higher scores mean more obsessive-compulsive personality traits.
The Emotion Regulation Questionnaire (ERQ) | 32 weeks
  A 10-item self-report questionnaire designed to measure adaptive and maladaptive strategies for emotion regulation. The adaptive subscale contains 6 questions and range between 6-42. Higher scores on this subscale mean more adaptive regulation strategies. The maladaptive subscale contains 4 questions and range between 4-28. Higher scores on this subscale mean more maladaptive regulation strategies.
Body mass index (BMI) | 32 weeks
  A statistical index using a person's weight and height to provide an estimate of body fat in people. A BMI of <18.5 indicates medically underweight. A BMI of 18.5 - 25 indicates normal weight. A BMI of >25 indicates overweight.
Client Satisfaction Questionnaire (CSQ-8) | 32 weeks
  An 8-item self-report questionnaire to measure patient satisfaction with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Sjögren, PhD, Principal Investigator — Umea University
Locations (1):
- Sundsvalls sjukhus, Lasarettsvagen 21, Sundsvall, Västernorrland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related link — https://pubmed.ncbi.nlm.nih.gov/24199611/
- See also: Related link — https://pubmed.ncbi.nlm.nih.gov/25346237/
- See also: Related link — https://pubmed.ncbi.nlm.nih.gov/33524917/